CLINICAL TRIAL: NCT01367210
Title: Switch to Darunavir/r + Maraviroc QD in Patients With R5 Tropism by Viral DNA Genotyping With Suppressed Viremia (GUSTA): a Multicenter, Open-label, Randomized Controlled Trial
Brief Title: Switch to Darunavir/r + Maraviroc Quaque Die in Patients With R5 Tropism by Viral DNA Genotyping (GUSTA)
Acronym: GUSTA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Because a higher rate of virological failures in study versus control arm.
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Simona Di Giambenedetto, Dr, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-023316-13
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: HIV Infection
Keywords: HIV; AIDS; Highly Active AntiRetroviral Therapy; Simplification; Maraviroc; Darunavir; Treatment experienced; Tropism
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MARAVIROC, DARUNAVIR/r (Experimental): Treatment simplification from a "standard" combined antiretroviral therapy including 3 drugs to Maraviroc plus Darunavir with Ritonavir. Treatment simplification from three-drugs- to two-drugs-based antiretroviral therapy
  Interventions: Drug: Maraviroc, Darunavir/r
- current ART with 3 drugs (Sham Comparator): Patients on HAART with three drugs and HIV RNA below 50 copies/mL
  Interventions: Drug: current antiretroviral therapy with 3 drugs

INTERVENTIONS:
Drug: Maraviroc, Darunavir/r — Maraviroc 300 mg Darunavir 800 mg Ritonavir 100 mg
  Arms: MARAVIROC, DARUNAVIR/r
Drug: current antiretroviral therapy with 3 drugs — To continue the assumption of previous HAART
  Arms: current ART with 3 drugs

SUMMARY:
Objectives of the study:

1. To verify the safety and the efficacy of the study treatment, defined as the persistent control of the virus' replication at 48 weeks after the simplification to maraviroc + darunavir with ritonavir in patients with R5 tropism by viral DNA genotyping.
2. To collect relevant information about the safety, the immunologic and the economic impact of this strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with the same regimen including 3 HAART from at least 4 months
* Aged 18 years or older
* Who gave informed consent to the participation to the study
* With at least two viral load < 50 copies/mL in two consecutive determinations at least 6 months apart (tolerance of two weeks)
* With CD4 cell count > 200 cells/μL and absence of any opportunistic infection or AIDS-related disease for at least one year prior to the screening.
* With R5 tropism by viral DNA genotyping (geno2pheno "clonal")
* With CD4 cell count nadir>50 cell/mmc or 100 cell/mmc if previous enfuvirtide or integrase inhibitors use

Exclusion Criteria:

* With at least one major or two minor mutation conferring resistance to darunavir reported in the update list of International AIDS Society - USA , in previous resistance test
* Previous D/M or X4 viral tropism
* Previous major clinical toxicities (grade >=3) to the proposed drugs of the study
* Pregnancy or breast feeding, desire of pregnancy in the short term
* Past exposure to Chemokine Receptor 5 antagonist
* HBsAg serostatus
* Liver cirrhosis of class C (Child-Pugh)
* Sulpha drug hypersensitivity
* The presence of major non AIDS-defining diseases that, in the opinion of the investigator, may compromise the retention of the patient in the study for the necessary follow-up period.
* Estimated glomerular filtration < 30 ml/min (cockroft-Gaut; MDRD formula if black-African or african-american) at screening visit
* Hypertransaminasemia of grade IV (more than 10 times the upper normal limit) at screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
proportion of patients with virological failure (two consecutive measures of HIV-RNA higher than 50 copies/mL or a single measure higher than 1000 copies/mL) within 48 weeks at per protocol analysis, with switch=failure | 48 weeks

SECONDARY OUTCOMES:
proportion of patients with virological failure (two consecutive measures of HIV-RNA higher than 50 copies/mL or a single measure higher than 1000 copies/mL) within 96 weeks at intention-to treat analysis with missing value=Failure | 96 weeks
Time to virological failure at survival analysis | 48 weeks
Proportion of patients with at failure X4 tropism viral tropism (RNA or DNA genotyping) | 48 weeks
Evolution of CD4 cell- cluster of differentiation 4 cell count during the 96 weeks | 96 weeks
Evolution of adherence and quality of life after 24, 48 and 96 weeks | 96 weeks
Evolution of maraviroc, darunavir, ritonavir plasma concentrations during the 96 weeks | 96 weeks
Evolution of metabolic parameters at 96 weeks | 96 weeks
Change of the results of neurocognitive tests at 48 and 96 weeks | 96 weeks
Modification of bone density and subcutaneous fat at 48 and 96 weeks | 96 weeks
Modification of Intima-Media Thickness and Flow Mediated Dilation at 48 and 96 weeks | 96 weeks
Economic impact of Darunavir/ritonavir+ Maraviroc versus Highly Active Antiretroviral Therapy | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Luca, Prof, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy